CLINICAL TRIAL: NCT06614296
Title: Factors and Experiences Associated with Unscheduled Hospital Readmission After Crenel Lateral Interbody Fusion
Brief Title: Unscheduled Hospital Readmission After Crenel Lateral Interbody Fusion
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0165
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Spine Degeneration
Keywords: Spine Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Unscheduled readimission: Unscheduled readimission after CLIF
  Interventions: Procedure: Crenel lateral interbody fusion plus second stage surgery
- Scheduled readimission: Scheduled readimission after CLIF
  Interventions: Procedure: Crenel Lateral Interbody Fusion

INTERVENTIONS:
Procedure: Crenel Lateral Interbody Fusion — The Crenel Lateral Interbody Fusion (CLIF) is a surgical technique developed by the Department of Spine Surgery at the Second Affiliated Hospital of Zhejiang University School of Medicine. Building on the traditional Lateral Lumbar Interbody Fusion technique, this series of technical improvements overcomes the shortcomings of previous surgical methods, enhancing the safety, operability, and effectiveness of the surgery while reducing complications.
  Other Names: Lateral Lumbar Interbody Fusion
  Groups: Scheduled readimission
Procedure: Crenel lateral interbody fusion plus second stage surgery — The patient was first admitted to undergo CLIF surgery and was discharged after the operation. The patient will return to the hospital for a second surgery at the scheduled time.
  Groups: Unscheduled readimission

SUMMARY:
The goal of this observational study is to learn about the readmission related to Crenel Lateral Interbody Fusion (CLIF). The main question it aims to answer is:

What are the risk factors for readmission after CLIF surgery?

ELIGIBILITY:
Inclusion Criteria:

* Patients with spinal degeneration undergoing CLIF surgery

Exclusion Criteria:

* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (>18 years old) with spinal degeneration undergoing CLIF surgery, including both unscheduled and scheduled readmissions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Unscheduled readmission | 1 year
  Unscheduled readmission refers to a patient who was unplanned or unexpected return to the hospital after CLIF discharged from a previous hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol